CLINICAL TRIAL: NCT01509716
Title: Assessing Perceived Versus Actual Knowledge and Quality of Life in Pre-Dialysis CKD Patients
Brief Title: Assessing Perceived Versus Actual Knowledge and Quality of Life in Pre-Dialysis Chronic Kidney Disease (CKD) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Priscilla How, Pharm.D., BCPS, Assistant Professor, National University of Singapore
Other Study IDs: DSRB Domain E/2011/02008
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease Stage 3; Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
Keywords: Predialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Aims: The investigators' primary objective is to assess both perceived and actual disease knowledge in local pre-dialysis Chronic Kidney Disease (CKD) patients. The investigators hypothesize that actual disease knowledge is poorer than perceived. As the secondary objectives, the investigators will also assess the HRQoL and examine the association between level of knowledge and HRQoL in pre-dialysis CKD patients. The investigators hypothesize that HRQoL of pre-dialysis CKD patients is poorer than that of the general population while pre-dialysis CKD patients with greater disease knowledge have a better HRQoL than those with poorer knowledge.

Methodology: A survey was developed to assess both perceived and actual knowledge on five aspects - general knowledge, nephrotoxic medications, diet restrictions, symptoms of CKD and its complications and renal replacement therapy (RRT) options. For the assessment of HRQoL, the following questionnaires will be used - Kidney Disease Quality of Life-Short Form (KDQOL-SF) version 1.3, EuroQoL 5 Dimensions (EQ-5D), Family Functioning Measure (FFM), and Oslo-3 Social Support Scale (OSS-3). All study questionnaires will be provided in 3 main languages - English, Chinese and Malay. A standardized data collection form was developed to retrospectively collect demographic and clinical information from the patients' electronic medical records and patient charts. Descriptive statistics will be used to report all results.

ELIGIBILITY:
Inclusion Criteria:

* patients at least 21 years of age,
* able to read English, Chinese or Malay,
* have stage 3 to 5 CKD as identified from their medical records, but are not receiving dialysis.

Exclusion Criteria:

* patients who do not consent,
* have already been started on dialysis,
* are cognitively impaired as assessed by the recruiter or unable to fill up questionnaires on their own.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Predialysis patients with stage 3-5 chronic kidney disease patients seen in outpatient renal clinic in National University Hospital, Singapore
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore